CLINICAL TRIAL: NCT00333346
Title: Tramadol iv. : Influence of Dose and Dose Intervals on Therapeutic Accuracy and Side Effects When Used for Postoperative Pain Relief in Ambulatory Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Michel Struys, University Hospital Ghent
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006/195
Record Dates: First submitted 2006-06-02; First posted 2006-06-05 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-08

CONDITIONS: Ambulatory Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Administration of tramadol intravenously

SUMMARY:
The aim of this study is to compare the administration of 1 unit dose of 100 mg tramadol intravenously versus multiple smaller dosages of tramadol during the first 6 hours post-operatively and to investigate the time course and accuracy of pain relief versus the onset and duration of side-effects.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II female or male patients
* Aged 18-70 years
* Scheduled for ambulatory surgery requiring postoperative pain medication.

Exclusion Criteria:

* Weight less than 70% or more than 130% of ideal body weight
* Neurological disorder
* Recent use of psycho-active medication, including alcohol
* Patients suffering from chronic pain receiving pre-operative pain medication including NSAID's
* Use of chronic anti-emetic medication, use of chronic corticoid therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Time course of pain relief
Accuracy of pain relief
Onset of side-effects
Duration of side-effects

CONTACTS AND LOCATIONS:
Overall Officials: Michel Struys, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be